CLINICAL TRIAL: NCT02414412
Title: Immunity Improvement Effect of Ulmus Macrocarpa Water Extract in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Collaborators: Bio Port Korea Inc. (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 022014031
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Ulmus macrocarpa water extract; immunity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ulmus (Active Comparator): Ulmus macrocarpa water extract 250mg orally 2 times a day for 4 weeks
  Interventions: Dietary Supplement: Ulmus macrocarpa water extract
- Placebo (Placebo Comparator): placebo 250mg orally 2 times a day for 4 weeks
  Interventions: Dietary Supplement: Ulmus macrocarpa water extract

INTERVENTIONS:
Dietary Supplement: Ulmus macrocarpa water extract

SUMMARY:
This randomized, placebo-controlled, double-blind study evaluates the efficacy and tolerability of Ulmus macrocarpa water extract for immunity improvement in relatively healthy adults. 58 subjects received 500 mg of Ulmus macrocarpa water extract per day or a placebo for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* subject has peripheral white blood cells between 4,000/Ul and 8,000/Ul

Exclusion Criteria:

* History of renal disease
* History of diabetes mellitus
* History of immune disease

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
serum natural killer cell activity | 1 month

SECONDARY OUTCOMES:
peripheral white blood cell | 1 month
serum tumor necrosis factor-alpha level | 1 month
serum interferon-gamma | 1 month
serum interleukins(1betta, 2,4,8,10, and 12) | 1 month

REFERENCES:
- [Derived] Cho AR, Lee SY, Cho YH, Kim CM, Kim SG. Effects of 4-Week Intervention with Ulmus macrocarpa Hance Extract on Immune Function Biomarkers in Healthy Adults: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2018 Feb 25;2018:5690816. doi: 10.1155/2018/5690816. eCollection 2018. PMID 29681977